CLINICAL TRIAL: NCT00703547
Title: A Single Blind, Randomized, Placebo Controlled, Crossover Study to Investigate the Safety, Tolerability and Pharmacokinetics of Single Oral Escalating Doses of GSK586529 in Healthy Volunteers
Brief Title: A First Time in Human Study of GSK586529 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Prevention
Other Study IDs: CRZ107432
Record Dates: First submitted 2008-04-14; First posted 2008-06-23 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Depressive Disorder and Anxiety Disorders
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects receiving treatment in cohort 1 (Experimental): Subjects will receive one of the following sequences; ABDF,BADF, BDAF or BDFA (A=Placebo, B= GSK586529 dose 1 (3 milligrams), D = GSK586529 dose 3, F = GSK586529 dose 5).
  Interventions: Drug: GSK586529 capsules; Drug: GSK586529 tablets; Drug: Placebo
- Subjects receiving treatment in cohort 2 (Experimental): Subjects will receive one of the following sequences; ACEG,CAEG, CEAG or CEGA (A = Placebo, C= GSK586529 dose 2, E = GSK586529 dose 4, G = GSK586529 dose 6)
  Interventions: Drug: GSK586529 capsules; Drug: GSK586529 tablets; Drug: Placebo

INTERVENTIONS:
Drug: GSK586529 capsules — GSK586529 will be provided as white gelatin capsule with a dose of 3 milligrams.
Drug: GSK586529 tablets — GSK586529 will be provided as a yellow film-coated tablets for oral administration at three different strengths 10 milligrams, 60 milligrams and 120 milligrams.
Drug: Placebo — Placebo tablets and capsules will be provided to subjects.

SUMMARY:
A single blind, randomized, placebo-controlled, crossover study in twenty four healthy male subjects. Subjects will be divided into two cohorts with alternate panel design. The study is investigating the safety, tolerability and pharmacokinetics of single oral escalating doses of GSK586529.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 18-45 years, inclusive.
* Healthy subjects, defined as individuals who are free from clinically significant illness or disease as determined by their (and familial) medical and psychiatric history, physical examination, laboratory studies, and other tests.
* Body weight >/= 50 kg (110 lbs) and BMI within the range 18.5-29.9 kg/m2 inclusive.
* Demonstrates no evidence of active disease, physical or mental impairment.
* Self-administered Beck Depression Inventory II scale total score no greater than 9, and suicide question score of zero.
* Non-smoker (abstinence from smoking for at least 6 months before the start of the study).
* Normal electrocardiogram (subjects must have no clinically significant abnormalities on a 12-lead ECG and a 24 hour Holter ECG).
* Read, comprehend, and write English at a sufficient level to complete study-related materials.

Exclusion Criteria:

* As a result of any of the medical interview, physical examination, evaluation of mental state and psychiatric history or screening investigations the physician responsible considers the subject unfit for the study.
* The subject has a positive pre-study drug/alcohol screen.
* A positive pre-study HIV, Hepatitis B surface antigen or positive Hepatitis C antibody
* The subject has a history of psychiatric illness.
* Any history of suicidal attempts or behavior.
* Abuse of alcohol defined as an average weekly intake of greater than 21 units or an average daily intake of greater than three units..
* Consumption of grapefruit juice or grapefruit within 14 days prior to the first dose of study medication.
* Any subject who is not prepared to eat the standard meals provided by the clinic or is a vegetarian.
* Any history of an endocrine disorder including, but not limited to, diabetes or disorders of the hypothalamus, pituitary, adrenal, or thyroid glands, or gonadal disorder or dysfunction of the reproductive organs.
* Clinically significant abnormal; total and free testosterone, LH, FSH, ACTH or cortisol, or TSH or T4 values at screening/baseline
* LFTs elevated
* Any other clinically significant laboratory abnormality
* The subject has a screening ECG with parameters outside ranges defined in the protocol will also be excluded.
* History of long QT syndrome (personal or family) or other cardiac conduction disorder, or other clinically significant cardiac disease.
* The subject has received an investigational drug or participated in any other research trial within 3 months or 5 half-lives, or twice the duration of the biological effect of any drug(whichever is longer) prior to the first dose of study medication.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John'sWort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* History or presence of allergy to the study drug or drugs of this class, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* Donation of more than 500 mL blood within the 3 months before dosing.
* An unwillingness of male subjects to abstain from sexual intercourse with pregnant or lactating women from the time of the first dose of study medication until 90 days following administration of the last dose of study medication
* An unwillingness of the male subject to use a condom/spermicide in addition to having their female partner use another form of contraception if the woman could become pregnant from the time of the first dose of study medication until 90 days following administration of the last dose of study medication.
* Current or recent (within one year) gastrointestinal disease; a history of malabsorption, esophageal reflux, peptic ulcer disease, irritable bowel syndrome; frequent (more than once a week) occurrence of heartburn; or any surgical intervention (e.g., cholecysectomy) which would be expected to influence the absorption of drugs.
* Average daily caffeine intake equivalent to > 4 cups of coffee or > 6 cups of tea.
* A semi-supine systolic blood pressure less than 90mmHg or greater than 140mmHg or a semi-supine diastolic blood pressure of less than 60mmHg or greater than 90mmHg; or a radial pulse rate less than 40bpm or more than 90bpm.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2008-01-28 (Actual); Primary Completion 2008-04-11 (Actual); Study Completion 2008-04-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | Pre-dose, 30 minutes, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post-dose

SECONDARY OUTCOMES:
Blood levels of GSK586529 to determine pharmacokinetic parameters | Pre-dose, 30 minutes, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post-dose
Urinary recovery of GSK586529 | Pre-dose, 0-6, 6-12, 12-24, 24-48, 48-72 and 72-96 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- See also: Results for study CRZ107432 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/CRZ107432?search=study&study_ids=CRZ107432#rs